CLINICAL TRIAL: NCT02640118
Title: The Impact of Lixisenatide on Postprandial Glucose Tolerance in Pancreatectomised Subjects -a Delineation of Extrapancreatic Effects
Brief Title: The Impact of Lixisenatide on Postprandial Glucose Tolerance in Pancreatectomised Subjects
Acronym: Px-Lixi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Principal Investigator, Filip Krag Knop, Associated Professor, MD, P.h.D., University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15004078
Record Dates: First submitted 2015-12-11; First posted 2015-12-28 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Diabetes After Total Pancreatectomy
MeSH Terms: interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pancreatectomised + Lixisenatide (Active Comparator): During the experimental day the patient will ingest a standardized liquid meal (200 ml containing 1,650 kJ (394 kcal): carbohydrate 50%, protein 15%, fat 35%, consisting of glucose (48.4 g + 1.6 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol).
  Before the meal a Lixisenatide-injection will be given subcutaneously
  Interventions: Drug: Lixisenatide; Other: Standardized liquid meal
- Pancreatectomized + lixisenatide-placebo (Placebo Comparator): During the experimental day the patient will ingest a standardized liquid meal (200 ml containing 1,650 kJ (394 kcal): carbohydrate 50%, protein 15%, fat 35%, consisting of glucose (48.4 g + 1.6 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol).
  Before the meal a placebo-injection will be given subcutaneously.
  Interventions: Drug: Lixisenatide-Placebo; Other: Standardized liquid meal
- Healthy + Lixisenatide (Active Comparator): During the experimental day the subject will ingest a standardized liquid meal (200 ml containing 1,650 kJ (394 kcal): carbohydrate 50%, protein 15%, fat 35%, consisting of glucose (48.4 g + 1.6 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol).
  Before the meal a Lixisenatide-injection will be given subcutaneously
  Interventions: Drug: Lixisenatide; Other: Standardized liquid meal
- Healthy + lixisenatide-placebo (Placebo Comparator): During the experimental day the subject will ingest a standardized liquid meal (200 ml containing 1,650 kJ (394 kcal): carbohydrate 50%, protein 15%, fat 35%, consisting of glucose (48.4 g + 1.6 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol).
  Before the meal a placebo-injection will be given subcutaneously
  Interventions: Drug: Lixisenatide-Placebo; Other: Standardized liquid meal

INTERVENTIONS:
Drug: Lixisenatide — single injection of 20 µg lixisenatide subcutaneously
  Other Names: Lyxumia
  Arms: Healthy + Lixisenatide; Pancreatectomised + Lixisenatide
Drug: Lixisenatide-Placebo
  Arms: Healthy + lixisenatide-placebo; Pancreatectomized + lixisenatide-placebo
Other: Standardized liquid meal — standardized liquid meal (200 ml containing 1,650 kJ (394 kcal): carbohydrate 50%, protein 15%, fat 35%, consisting of glucose (48.4 g + 1.6 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol).

SUMMARY:
Postprandial glucose (PPG) excursions are not only determined by insulin-mediated glucose disposal and endogenous glucose production (regulated by insulin and glucagon); also the rate of gastric emptying constitutes an important determinant of PPG levels 1. The short-acting glucagon-like peptide-1 (GLP-1) receptor agonist lixisenatide is used in the treatment of type 2 diabetes. It increases glucose-dependent insulin secretion, suppresses glucagon secretion and reduces gastric emptying of meals 2. These three mechanisms most likely constitute the weightiest mechanisms behind the potent impact of lixisenatide on exaggerated PPG excursions in patients with type 2 diabetes - which often are normalised during lixisenatide treatment 3. However, the separate impact of lixisenatide-induced reduction of gastric emptying (independently of the pancreatic effects) has been difficult to determine. Importantly, treatment with lixisenatide also decreases appetite and food intake and may, like native GLP-1, increase energy expenditure 4. So far an exact demarcation of the pancreatic and extrapancreatic effects of lixisenatide in humans remains to be established.

The present project serves to determine whether effects of lixisenatide on gastric emptying, appetite, food intake and resting energy expenditure are dependent on the endocrine pancreas.

The study is a randomised, placebo-controlled, double-blinded, cross-over study.

12 healthy persons and 12 pancreatectomized patients (i.e. patients who have had their pancreata removed due to pancreatic cancer or severe chronic pancreatitis) will be subjected to two experimental days on which they will undergo a liquid meal test followed by a fasting period and finished off with an ad libitum meal with lixisenatide and placebo, respectively.

ELIGIBILITY:
Inclusion criteria Pancreatectomised patients

* Caucasians above 18 years of age who have undergone total pancreatectomy
* Normal haemoglobin
* Informed consent Healthy subjects
* Normal fasting plasma glucose (FPG) and normal HbA1C (according to the World Health Organization (WHO) criteria)
* Normal haemoglobin
* Age above 18 years
* Informed consent

Exclusion criteria Pancreatectomised patients

* Inflammatory bowel disease
* Operation within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Ostomy
* Nephropathy (serum creatinine >150 µM and/or albuminuria)
* Severe liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigator feels would interfere with trial participation Healthy subjects
* Diabetes mellitus (DM)
* Prediabetes (impaired glucose tolerance and/or impaired FPG)
* First degree relatives with DM
* Inflammatory bowel disease
* Intestinal resection and/or ostomy
* Nephropathy (serum creatinine >150 µM and/or albuminuria
* Liver disease (ALAT and/or serum ASAT >2×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
PPG excursions measured as incremental area under curve (iAUC) | -120,-45,-30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes

SECONDARY OUTCOMES:
differences in gastric emptying, measurement of s-paracetamol | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
  measurement of time to peak and incremental area under the curve (iAUC)
food intake and appetite | at time 0,30,60,90,120,150,180 minutes
  assessed by a visual analogue scale (VAS)
resting energy expenditure (REE) | -90,30,150 minutes
  measured by calorimetry
p-glucose mmol/L | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
p-C-peptide pmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
glucagon, gastrin, cholecystokinin, GIP, GLP-1, oxyntomodulin | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Assoc. Prof., Principal Investigator — Center for Diabetes Research, Gentofte Hospital, Kildegaardsvej 28, 2900 Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Juel CTB, Lund A, Andersen MM, Hansen CP, Storkholm JH, Rehfeld JF, van Hall G, Hartmann B, Wewer Albrechtsen NJ, Holst JJ, Vilsboll T, Knop FK. The GLP-1 receptor agonist lixisenatide reduces postprandial glucose in patients with diabetes secondary to total pancreatectomy: a randomised, placebo-controlled, double-blinded crossover trial. Diabetologia. 2020 Jul;63(7):1285-1298. doi: 10.1007/s00125-020-05158-9. Epub 2020 May 11. PMID 32394228